CLINICAL TRIAL: NCT00409669
Title: Study to Compare the Accuracy and Variability of the Barraquer Tonometer With Other Methods of Tonometry
Brief Title: Intraocular Pressure Accuracy and Variability of the Barraquer Tonometer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Barnes Retina Institute (Other)
Responsible Party: Arghavan Almony, M.d., Barnes Retina Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BRI 06-0987
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Elevated Intraocular Pressure
Keywords: Barraquer tonometer; Intraocular pressure; Tonometry
MeSH Terms: conditions — Ocular Hypertension

INTERVENTIONS:
Device: Barraquer tonometer — barraquer tonometer

SUMMARY:
To determine if the Barraquer tonometer provides an accurate and reliable measurement of intraocular pressure. The Barraquer tonometer is a device used to safely and painlessly measure intraocular pressure.

DETAILED DESCRIPTION:
Intraocular pressure will be checked using four different methods of tonometry. These four methods will include Tonopen, Goldmann applanation tonometry, Schiotz tonometry, and Barraquer tonometer. The data will then be compared to determine the reliability and accuracy of the Barraquer tonometer.

ELIGIBILITY:
Inclusion Criteria:

1. All patients of Barnes Retina Institute who are scheduled to undergo vitreoretinal surgery.
2. All patients scheduled for routine eye examination at the Washington University Eye Clinic or Barnes Jewish Eye Clinic.
3. All ages (patients seen at these locations are adult patients >18 years of age).

Exclusion Criteria:

1. Any patient who is seen in the outpatient clinics for an urgent or emergency ophthalmological issue.
2. Any patient who has a contraindication to routine, noninvasive methods of tonometry and/or pachymetry (ie corneal ulcer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-11 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Central corneal thickness as measured by pachymetry | at time of measurement
Intraocular pressure as measured by Schiotz tonometer | at time of measurement
Tonopen | at time of measurement
Barraquer tonometer | at time of measurement
and Perkins tonometer | at time of measurement

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Grand, MD, Principal Investigator — Washington University School of Medicine and Barnes Retina Institute
Locations (1):
- Washington University School of Medicine and Barnes Jewish Hospital, St Louis, Missouri, United States